CLINICAL TRIAL: NCT04371003
Title: Prospective Investigation of Oxidative Stress in West Nile Virus Infection
Acronym: PROWENI
Status: Withdrawn | Type: Observational
Why Stopped: Study proposal was not accepted for funding and therefore not further explored at this stage.
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Victor Babes Hospital, Bucharest, Romania (Unknown); Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Other Study IDs: ITM202005
Record Dates: First submitted 2020-04-09; First posted 2020-05-01 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: West Nile Virus; West Nile Fever; West Nile Fever Encephalitis; West Nile Fever Meningitis; West Nile Meningitis; West Nile Virus Meningoencephalitis; West Nile Fever Meningoencephalitis; West Nile Fever With Neurologic Manifestation; Oxidative Stress
Keywords: Genome sequencing; composite diagnosis
MeSH Terms: conditions — West Nile Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- WNND: 40 subject with West-Nile Neuroinvasive Disease will be recruited
- WNF: 40 subject with West-Nile Fever will be recruited
- controls: 20 control will be recruited. These controls will be aged matched to the cases.

SUMMARY:
The investigator hypothesizes that oxidative stress responses to West Nile virus infection in the central nervous system determine the severity of infection and the long-term neurological, neuropsychological and functional sequelae of West Nile Neuroinvasive Disease.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent. If the clinical condition of the patient does not permit giving consent, informed consent will be obtained from the next of kin.
* Age 18 years or older
* for active cases: positive anti-WNV IGM antibodies in serum (or IgG in CSF if applicable)
* for active cases: presentation within (maximum) 7days of symptom onset
* for healthy controls: anti-WNV antibody naive (IgM and IgG in serum). The group of healthy controls will be selected to have an age similar distribution to the cases.

Exclusion Criteria:

* Evidence of active systemic infection in 3 months prior to recruitment
* Evidence of systemic inflammatory illness
* Clinical signs of neurodegenerative or neurologic disease other than WNND
* Pregnancy
* Active malignancy
* History of drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be recruited from VBH emergency and outpatient departments in Bucharest, Romania, from the onset of the WNV transmission season in 2020 until November 2023. The incidence of WNV and WNND in South-Eastern Romania was 0.5 per 100,000 inhabitants in 2016, and has been increasing steadily 35. Romania reported 277 WNND cases with 43 deaths in 2018, and 66 WNND cases with 8 deaths in 2019 3. VBH is a tertiary care facility that serves a population of 3 million people (15% of Romania's population). Its catchment area covers more than 80% of the territories in Romania that reported WNV transmission and has in recent years been the largest single medical center to care for WNV infected patients.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure the redox status | at recruitment, 10 days post-symptom onset and 20 days post symtom onset.
  A multiparameter indexes of oxidative stress will be calculated to measure and summarize the redox status in cases and age matched controls. Association between the redox status and clinical, neuropsychological and radiological outcomes will be investigated. We will also examine the relative sensitivity of separate biomarkers of oxidative stress and autophagy as clinical predictors of WNV infection severity.
Assessment of Neurologic deficits | At recruitment, month 3 and month 12
  As part of the descriptive analysis of biomarkers of disease severity and to study to neurologic sequelae of WNV infection. Will be assessed: specifically assessments of cranial nerves II- XII, motor strength in upper and lower extremities, sensory testing for pinprick and vibration, deep tendon reflexes, gait, coordination, and movement abnormalities
Neuropsychologic performance | 20 days post-symtom onset, month 3 and month 12
  Study the neuropsychologic sequelae of WNV infection during a 12-month followup period in following key domains: Attention, Memory, Executive Function, Emotion & Social Cognition, Psychomotor Speed
Longitudinal assessment of functional status Study the neurologic and neuropsychologic sequelae of WNV infection during a 12-month followup period. | at recruitment, month 3 and month 12
  ECOG/WHO PS during a 12-month followup.
MRI abnormalities | at recruitment, month 3 and month 12
  Part of descriptive analysis of clinical markers of disease severity
Brain iron content | at recruitment, month 3 and month 12
  Part of the descriptive analysis of clinical markers of disease severity: Qualitative analysis per neuroanatomical region by iron-sensitive MRI sequence (SWI)
Ophthalmological abnormalities | at recruitment, with a follow-up of clinically indicated.
  As part of the descriptive analysis of clinical markers of disease severity ophthalmologic abnormalities will be assessed by slit lamp examination
serum S100b concentration | at recruitment, 10 days post symptom onset and 20 days post symptom onset
  As part of the descriptive analysis of clinical markers of disease severity S100b concentration will be measured to asses the Blood-Brain barrier integrity
serum NSE concentration | at recruitment, 10 days post symptom onset and 20 days post symptom onset
  As part of the descriptive analysis of clinical markers of disease severity NSE concentration will be measured to asses the Blood-Brain barrier integrity

SECONDARY OUTCOMES:
Analysis of laboratory performance characteristics (e.g. sensitivity) of WNV-specific RT-PCR and viral isolation in clinical samples, compared to composite diagnosis of WNV infection | 20 days
  Confirmed WNV infection is defined as one or more of following criteria:
  1. Seroconversion of anti-WNV IgG antibodies (Indirect immunofluorescence testing (IIFT) Flavivirus 2, Euroimmun®, Lübeck, Germany) in convalescent serum (20 days after symptom onset) (all participants)
  2. 4-fold increase of anti-WNV IgG antibodies in convalescent serum, compared to the screening sample (IIFT).
  3. Anti-WNV IgM antibody detection (ELISA) in CSF* (at VBH) (*CSF sampled only when clinically indicated).
  4. Positive WNV-specific RT-PCR result in serum, urine or CSF in samples obtained at screening.
  5. Virus isolation by outgrowth assay in samples obtained at screening
Description of molecular epidemiology of infecting WNV strain(s) and viral outgrowth diagnostic performance. | 20 days
  The time frame for WNV detection after symptom onset by real-time reverse transcriptase polymerase chain reaction (RT-PCR) or virus isolation by outgrowth from blood or CSF is limited by the fast decline of circulating virus. Because the WNV RNA detection window in urine can be longer (up to 14 days), RT-PCR will be performed on all clinical samples at recruitment. The target sequences are a conserved region in the 5'UTR region and part of the capsid gene of WNV and detects both lineage 1 and 2 WNV. WNV has been successfully isolated from urine, in approx. 40% of samples obtained within 8 days of symptom onset. WNV isolation will be attempted in low-passage Vero E6 cells and BHK21 cells from urine samples with a high WNV RNA load (Cycle threshold (Ct)- values <30).
Identification of potential genetic signatures that correlate with virulence (neuro-invasion and morbidity) in our cohort. | 20 days
  Whole genome sequencing (WGS) will be performed on a subset of RT-PCR positive serum, urine and CSF samples. This will allow us to investigate the temporal and spatial compartmentalization of the West Nile lineages in Romania as well as expand our understanding of genetic compartmentalization within hosts (urine, serum, CSF). In addition, the obtained isolates will be sequenced (from the viral outgrowth assay) to assess potential adaptations the virus undergoes during isolation. Finally, in a genome wide association study, the obtained viral sequences will be compared with the prospectively collected clinical data, to identify potential genetic signatures that correlate with virulence, neuroinvasion and morbidity. Our data will be compared to existing data on genetic determinants of virulence such as the presence of a glycosylation site in the E protein, substitutions in non-structural proteins 3, 4B or 5, or variation in the 3' noncoding region.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Vercauteren, Principal Investigator — Institute of Tropical Medicine Antwerp; Nina Hermans, Principal Investigator — Universiteit Antwerpen; Corneliu Popescu, Principal Investigator — Victor Babes Hospital, Bucharest
Locations (1):
- Victor Babes Hospital, Bucharest, Romania